CLINICAL TRIAL: NCT06440434
Title: Effects of Morningness on Night Split Shift Performance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Ståle Pallesen, Professor, University of Bergen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M3447
Record Dates: First submitted 2024-05-14; First posted 2024-06-03 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Shift-work Disorder

STUDY DESIGN:
Intervention Model Description: A 2 (midnight-4am vs.4am-8am) within factor x 2 (below vs. above median on morningness) between factor experimental design
Masking Description: Randomly allocated to order of night shifts (midnight-4am vs.4am-8am)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early night shift (midnight-4am) (Active Comparator)
  Interventions: Behavioral: Time of night shift
- Late night shift (4am - 8am) (Active Comparator)
  Interventions: Behavioral: Time of night shift

INTERVENTIONS:
Behavioral: Time of night shift — Early vs. late night split night shift

SUMMARY:
The goal is to investigate if the morningness-eveningness dimension mediates sleep and function on spilt night shifts (midnight-4am and 4am-8am).

Does those with high score of morningness function relatively better on the last compared to the first split shift?

Participants will:

Record their sleep from 2 days prior to 2 days following the split shift During the shifts complete questionnaires assessing mood, sleepiness and perceived performance as well as complete cognitive tests: Psychomotor vigilance test, digit symbol substitution test, working memory scanning test, reversal learning test, and visual search test

DETAILED DESCRIPTION:
A sample of 28 students will be recruited and exposed to two conditions in a randomized, controlled, crossover study. They will be assessed with subjective (sleep diary) and objective sleep measures (sleep radar) for 2 days before the night shift, during the night shift and 2 days following the night shift. The simulated night shifts will last from midnight to 8am and will be divided into two halves (midnight-4am and 4am-8am), denoted as split-shift, and for each participant separated by at least 1 week. Based on the Horne-Östberg Morningness-Eveningness Questionnaire (median spilt) two groups are created, from which participants will be randomized to the two orders of the spilt-shift.

Each hour on each shift the participants will complete: Positive and Negative Affect Schedule (PANAS), Karolinska Sleepiness Scale, perceived performance and the following cognitive tests: Psychomotor vigilance test, Digit symbol substitution test, Working memory scanning test, Reversal learning test, and Visual search test.

Data will be analyzed with linear mixed models with three fixed factors: Group (low vs. high morningness), shift (midnight-4am vs. 4am-8am), and hour and one random factor (participant).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* no incorrectable vision problems

Exclusion Criteria:

* regular use of sleep medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | Total sleep time between 6pm day before shift start to 6pm the day the shift end for both early night shift (midnight-04am) and late night shift (04am-08am)
  Total sleep (sleep diary and radar). Higher values indicates more sleep
Psychomotor Vigilance Test (PVT) | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Reaction time (mean 1/RT) and number of lapses (RTs≥500 ms). For mean 1/RT higher values are associated with best performance, on lapses higher values are associated with worst performance
Karolinska Sleepiness Scale (KSS) | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Assessment of state sleepiness, range 1-9 (higher scores indicate worse state)

SECONDARY OUTCOMES:
Sleep efficiency (percentage of time in bed one sleeps) | Between 6pm day before shift start to 6pm the day the shift end for both early night shift (midnight-04am) and late night shift (04am-08am)
  Sleep efficiency (diary and radar). Range from 0-100%. Higher scores indicate best state
Positive and Negative Affect Schedule (PANAS) | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Assessment of mood/affect. Range 10-50. On positive mood subscale higher scores indicate best state, on negative mood state, higher scores indicate worst state
Self-rated performance | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Self-rated performance on cognitive tests. Range 1-10. Higher scores indicate best performance rating
Digital Symbol Substitution Test | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Test where one match symbols to numbers as fast as possible. Range 0-100. Higher scores indicate best performance
Working Memory Scanning Test (probed recall) | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Test presenting list of words. Then words are presented and subjects decide if word was present or not in list presented. The accuracy and RTs for positive trials (where probe was present in list) will be used as dependent variables. Higher accuracy and lower reaction time are associated with best performance
Reversal Learning Test | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Test measuring the ability to differentiating between "go-stimuli" and "no-go stimuli" before and after reversal of go and no-go stimuli. Discriminability (hit rate/false alarm rate) and response bias before and after reversal are recorded. Higher discriminability indicates better performance, higher response bias indicate worse performance
Visual Search Test | Hourly during shifts (0:15am, 1:15am, 2:15am and 3:15am on early night shift; 4:15am, 5:15am, 6:15am and 7:15 am on late night shift)
  Multiple objects are presented, and from among them a target is identified. The task of the subject is finding the target. Outcomes are reaction time (RT) and accuracy. Lower reaction times and higher accuracy are associated with best performance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
If legel in terms of data protection regulations data will be shared